CLINICAL TRIAL: NCT02757261
Title: Evaluation of Muscle Activity, Bite Force and Salivary Cortisol in Children With Bruxism Before and After Laser Use of Low Power in Acupoints- Controlled Clinical Trial
Brief Title: Evaluation of Muscle Activity, Bite Force and Salivary Cortisol in Children With Bruxism
Acronym: Bruxism
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Monica Canuto Salgueiro, Monica Canuto Salgueiro, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.333.636
Record Dates: First submitted 2016-04-08; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Sleep Bruxism
Keywords: Bruxism; Child; Occlusal splint; Bite force; Acunpuncture; Laser; Muscle actvity; Salivary Cortisol
MeSH Terms: conditions — Sleep Bruxism; Bruxism | interventions — Lasers; Occlusal Splints

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Application of Low-level laser therapy. (Experimental): The intervention will be twelve sessions (two per week). Laser parameters: wavelength - 786.94 nm; conventional tip; energy density - 25 J/cm²; intensity - 1.675 mW/cm²; output power - 70 mW (0.070 W); and exposure time - 20 seconds per point. The point application method will be used with direct contact with the skin (spot beam of 0.04 cm²), following the protocol suggested by Carvalho et al.50 and Venezian et al.44 A potentiometer will be used to determine the mean power of the laser equipment to ensure the safety of the operator.
  Interventions: Device: Laser
- Treatment with Occlusal splint. (Experimental): The intervention will be a maxillary occlusal splint will be used on the maxilla with palatal and occlusal coverage. Following the protocol established by Hachmann et al., the children will only use the splint at night for two months, with weekly adjustments of a quarter turn.46
  Interventions: Device: Occlusal splint
- Placebo laser (Active Comparator): Placebo laser will be performed using the same equipment.
  Interventions: Device: Placebo laser
- Children without bruxism (No Intervention): Control group

INTERVENTIONS:
Device: Laser — Low-level laser therapy administrated to acupoints
  Arms: Application of Low-level laser therapy.
Device: Occlusal splint — Occlusal splint with expander
  Arms: Treatment with Occlusal splint.
Device: Placebo laser — Placebo laser (Low-level laser therapy administrated to acupoints)
  Arms: Placebo laser

SUMMARY:
Bruxism is a repetitive activity of the masticatory muscles characterized by grinding and/or clenching one's teeth or parafunctional movements of the mandible. The aim of the proposed controlled clinical trial is to evaluate muscle activity, bite force and salivary cortisol in children aged six to eight years with bruxism. The children will be randomly allocated to four groups, each with 19 participants: Group 1 will receive low-level laser therapy at acupuncture points; Group 2 will use an occlusal splint; Group 3 will receive placebo laser therapy; and Group 4 will be the control group without bruxism. Low-level laser (786.94 nm, 0.04 cm2, 70 mW and 20 s per points) will be applied directly on the skin at six acupuncture points on each side. The BTS TMJOINT electromyograph will be used to determine muscle activity and a digital gnathodynamometer will be used to measure bite force. Two saliva collections will be performed in the participant's home at 9 am and prior to going to sleep, with at least one hour of fasting and followed by oral hygiene with water. Evaluations will be performed before as well as one and six months after treatment. The findings will be computed and submitted to statistical analysis. Descriptive statistics will be used first for the determination of point estimates, precision and validation using analysis of variance (ANOVA) for the evaluation of residuals and parametric tests will be used for the determination of pre-treatment conditions. Interval estimates will be used for the variables of interest to determine the prevision of the estimates and perform comparisons. When necessary, transformation methods or non-parametric tests will be used in the data analysis. The chi-square test, Student's t-test and ANOVA will be employed, with the level of significance set at 5% (p < 0.05).

DETAILED DESCRIPTION:
The aim of the proposed study is to evaluate the electromyographic activity of the masseter, anterior temporal and trapezius muscles as well as bite force, occlusal contacts and salivary cortisol following the administration of low-level laser therapy at acupoints or occlusal splint usage in children with sleep bruxism.

A randomized, controlled, clinical trial is proposed, which will be conducted in compliance with the norms governing research involving human subjects, following approval from the Institutional Review Board of University Nove de Julho (Brazil) under process number 1.333.636. The participants and/or legal guardians will receive clarifications regarding the objectives and procedures and will sign a statement of informed consent.

Individuals making use of muscle relaxants, those with temporomandibular disorder and those currently undergoing another treatment for bruxism will be excluded from the study.

Male and female children aged six to eight years with no physical or psychiatric limitations that may compromise the proposed therapies will be included. All individuals will need to have the first molars in Angle Class I and be free of dental caries. A clinical examination of tooth wear and the reports of parents/caregivers regarding tooth clenching/grinding will be used for the diagnosis of bruxism, following the criteria established by the American Academy of Sleep Medicine1 and the use of a questionnaire adapted by Serra Negra (2014).

The participants will be randomly allocated to four groups. Evaluations will be performed before and after treatment. Muscle activity will be determined using the BTS TMJOINT® device; bite force will be determined using a gnathodynamometer and salivary cortisol will be measured.

The electrical activity resulting from the activity of the massester and anterior temporal muscles will be determined using the six-channel BTS TMJOINT electromyograph (BTS Engineering), with a bioelectric signal amplifier, wireless data transmission and disposable bipolar surface electrodes (Ag/AgCl - Medical Trace®) measuring 10 mm in diameter. The electromyographic (EMG) signal will be amplified with a gain of 2000 times and filtered within a frequency of 20 to 450 Hz. The impedance will be >1015 Ω//0.2 pF and the common rejection mode will be 60/10Hz 92 dB. The data will be digitized at 1000 frames per second using the BTS MYOLA® program.52 Surface EMG signals will be recorded in the right and left masseter and anterior temporal bundles with disposable surface electrodes (Ag/AgCl - Medical Trace®) measuring 10 mm in diameter attached over the belly of the muscle in the region of the greatest tonus (determined during maximum voluntary clenching). The positioning of each electrode will follow the recommendations of the Surface EMG for the Non-Invasive Assessment of Muscles.52 Bandage tape will used to secure the electrodes further, with care taken to avoid micro-movements. The inter-electrode distance will be 20 mm from center to center.Prior to attachment, the sites for the electrodes will be cleaned with a cotton ball soaked in alcohol to diminish impedance. A reference electrode (3 x 2 cm) coated with Lectron II conductive gel (Pharmaceutical Innovations®) will be attached to the left wrist of the volunteer to allow the recording of differential signals.

To standardize the EMG potentials of the four muscles analyzed with occlusal contacts, two strips of Parafilm M® (American National Can TM, Chicago, USA) folded into five parts (10 mm in thickness) will be positioned bilaterally over the mandibular first and second molars of each subject. The electrodes will transfer data to a portable device with a real-time display. The system will process and compare the data with a set of predefined models for the evaluation of muscle activity during specific tasks.52 The EMG signal will be amplified and digitized (gain of 150 x, peak-to-peak input of 28 ± 14 mV, resolution of 12 b, sampling frequency of 2230 Hz A/D and theoretical resolution of 16 IV) using a differential amplifier with a rejection rate of 105 dB in the range of 0 to 60 Hz, input impedance of 10 GX and low-pass analog filter with a band width of 0 to 580 HZ as well as a digital filter with a band width of 30 to 400 Hz. The signals will be recorded for subsequent analysis.

Maximum voluntary clenching (MVC) will be recorded for four seconds three times with a three-minute interval between readings. After five minutes of rest, EMG activity will be recorded for 15 seconds three times successively each under the following conditions: i) Resting position: the subject will be instructed to relax and maintain the maxillary and mandibular teeth out of contact; ii) maximum voluntary clenching (isometric): the subject will be instructed to clench as hard as possible; and iii) chewing (isotonic): the subject will be instructed to lightly and systematically bite down on the two strips of parafilm positioned bilaterally in time with a metronome calibrated at 60 beats per minute. A three-minute interval between readings will be given for the EMG signals recorded in the resting position and during chewing and a five-minute interval between readings will be used for MVC.

A point 2 cm to the side of the midpoint of a line between the posterior margin of the acromion and the seventh cervical vertebra will be used for the positioning of the electrodes on the descending fibers of the trapezius muscle. Prior to the reading, the participant will be instructed to remain seated in a chair, with bare shoulder and arm, back straight, knees flexed at 90º and feet apart for the collection of MVC. Two non-elastic straps attached to each side of the base of the chair will be used to resist the elevation of the shoulders during the MVC reading. The volunteer will be instructed to raise the shoulders with maximum force for five seconds. This procedure will be performed three times with a one-minute rest period between readings and the largest value of the three readings will be used for the normalization of the EMG data of the descending fibers of the trapezius muscles.

After a three-minute interval, the volunteer will be instructed to perform 90° abduction of both arms for 60 s with the elbows completely extended and the forearms in pronation with the palms of the hands turned toward the floor. To monitor the positioning of the shoulders, two flexible bars positioned horizontally at a distance of 8 cm between the arms will be used to provide feedback of the tactile position.

A clinical examination will be performed to determine the type of occlusion based on the Angle classification, which is the most practical, traditional method and considered the gold standard in the literature.56 This system is based on the anteroposterior relationships of the jaws.

Bite force will be measured using a digital gnathodynamometer (DMD, Kratos Equipamentos Industriais Ltda, Cotia, São Paulo, Brazil) adapted for oral conditions. Readings will be taken in the region of the first molars. The participants will receive instructions and previous training to become familiarized with the device. According to the specific literature, the vertical movement of the mandible in the age group analyzed ranges from 35 to 40 mm. The digital dynamometer adapted to oral conditions has a capacity of up to 100 Kgf and has two beams measuring approximately 10 mm in diameter to avoid muscle stretching and ensure that the vertical movement of the mandible does not affect the force employed.

Six readings will be performed (three on the right and three on the left side), alternating sides between readings. Each reading will last five seconds, with a one-minute rest period between readings. The evaluation will be performed prior to treatment, immediately after treatment and 30 days after treatment. The results will be computed and analyzed statistically.

A maxillary occlusal splint will be fabricated in colorless acrylic resin and used on the maxilla with palatal and occlusal coverage. Molds of the maxillary and mandibular arches will be made in alginate for the fabrication of plaster models with a semi-adjustable joint. The splint will first be fabricated with dental wax in two layers and adapted to the maxillary teeth. The splint will measure 3 mm in thickness and will have contact with all teeth in a centric relationship, distal occlusion of the posterior teeth in laterality and protrusion, avoiding interferences on the side of balance with the guide canine, extending in the vestibular to lingual direction enough to prevent perforation and increase resistance to impact. An expander will also be placed so that the splint can accompany craniofacial growth. Following the protocol established by Hachmann et al., the children will only use the splint at night for two months, with weekly adjustments of a quarter turn.46 Saliva will be collected on cotton swabs, which will be left in the mouth for two minutes. The cotton will then be placed into a centrifuge tube and the sample will be stored at -20° C until analysis.25 Salivary cortisol will be measured prior to therapy and on Day 50 to measure the degree of stress. Two collections will be performed in the home of the participant at 9 am and prior to going to sleep with at least one hour of fasting prior to the collection and will be followed with oral hygiene with water. The collection will be performed on a Sunday following the manufacturer's recommendations and will be delivered on the following Monday for analysis at University Nove de Julho (Brazil).

The child will be seated comfortably in a room without noise or sound interference, with the head positioned on the Frankfurt plane (parallel to the floor). The active tip of the laser will be covered with plastic wrap to avoid cross-contamination and for reasons of hygiene. The site to be irradiated will be previously cleaned with 70% alcohol. Twelve sessions will be performed (two per week). The following will be the laser parameters: wavelength - 786.94 nm; conventional tip; energy density - 25 J/cm²; intensity - 1.675 mW/cm²; output power - 70 mW (0.070 W); and exposure time - 20 seconds per point. The point application method will be used with direct contact with the skin (spot beam of 0.04 cm²), following the protocol. A potentiometer will be used to determine the mean power of the laser equipment to ensure the safety of the operator.

One group will receive active LLLT and one group will receive placebo LLLT over the following acupoints:

IG-4 (Hegu) - This point exerts a strong, direct influence on the eyes, ears, nose and mouth; this point is also used to calm the mind and alleviate anxiety; F-3 (Taichong) - This point exerts a profound calming effect on the mind, which is enhanced when combined with IG-4; VB-34 (Yanglingquan) - This point is important to the relaxation of the tendons whenever muscles contract; E-36 (Zusanli) - This point is indicated to treat irritability, depression, insomnia, tiredness, fatigue and headache; ID-19 (Ting gong) - This point is indicated for the treatment of problems in the region of the ear; BP-6 (Sanyinjiao) - This is one of the most important points, with a broad scope of action, including a strong calming effect on the mind, and is used to treat insomnia.

Placebo laser will be performed using the same equipment. For such, the device emits a red guide light and sound, but does not emit energy. After 30 days, the volunteers in the placebo group will receive complementary treatment for the control of bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children
* Aged six to eight years
* No physical or psychiatric limitations
* Need to have the first molars in Angle Class I
* Free of dental caries
* A clinical examination of tooth wear and the reports of parents/caregivers regarding tooth clenching/grinding will be used for the diagnosis of bruxism, following the criteria established by the American Academy of Sleep Medicine1 and the use of a questionnaire adapted by Serra Negra (2014).

Exclusion Criteria:

* Use of muscle relaxants
* Temporomandibular disorder
* Currently undergoing another treatment

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in ELECTROMYOGRAPHIC EVALUATION OF MASTICATORY AND TRAPEZIUS MUSCLES | Before and after treatment and follow up 1 month and 6 months
  six-channel BTS TMJOINT electromyograph (BTS Engineering)
Change in Bite force | Before and after treatment and follow up 1 month and 6 months
  Bite force will be measured using a digital gnathodynamometer (DMD, Kratos Equipamentos Industriais Ltda, Cotia, São Paulo, Brazil) adapted for oral conditions
Change in Salivary cortisol | Before and after treatment and follow up 1 month and 6 months
  Saliva will be collected on cotton swabs, which will be left in the mouth for two minutes. The cotton will then be placed into a centrifuge tube and the sample will be stored at -20° C until analysis.25 Salivary cortisol will be measured prior to therapy and on Day 50 to measure the degree of stress. Two collections will be performed in the home of the participant at 9 am and prior to going to sleep with at least one hour of fasting prior to the collection and will be followed with oral hygiene with water. The collection will be performed on a Sunday following the manufacturer's recommendations and will be delivered on the following Monday for analysis at University Nove de Julho (Brazil).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salgueiro MDCC, Bortoletto CC, Horliana ACR, Mota ACC, Motta LJ, Motta PB, MesquitaFerrari RA, Fernandes KPS, Bussadori SK. Evaluation of muscle activity, bite force and salivary cortisol in children with bruxism before and after low level laser applied to acupoints: study protocol for a randomised controlled trial. BMC Complement Altern Med. 2017 Aug 8;17(1):391. doi: 10.1186/s12906-017-1905-y. PMID 28789647